CLINICAL TRIAL: NCT02606253
Title: Comparison of Oral Thiazides vs Intravenous Thiazides vs Tolvaptan in Combination With Loop Diuretics for Diuretic Resistant Decompensated Heart Failure
Brief Title: Comparison of Oral or Intravenous Thiazides vs Tolvaptan in Diuretic Resistant Decompensated Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Zachary L. Cox, Associate Professor, Lipscomb University College of Pharmacy, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VU-IRB-TBD
Record Dates: First submitted 2015-11-11; First posted 2015-11-17 (Estimated); Results first posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-10

CONDITIONS: Heart Failure
Keywords: loop diuretics; thiazide diuretics; vasopressin antagonists; diuretic resistance; heart failure
MeSH Terms: conditions — Heart Failure | interventions — Tolvaptan; Chlorothiazide; Metolazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Metolazone (Active Comparator): Metolazone 5mg tablet orally twice daily for 48 hours.
  Interventions: Drug: Metolazone
- Chlorothiazide (Experimental): Chlorothiazide 500mg intravenous infusion over 30 minutes twice daily for 48 hours
  Interventions: Drug: Chlorothiazide
- Tolvaptan (Experimental): Tolvaptan 30mg tablet orally once daily for 48 hours
  Interventions: Drug: tolvaptan

INTERVENTIONS:
Drug: tolvaptan — Tolvaptan (Samsca) is a vasopressin 2 receptor antagonist that works in the collecting duct of the nephron to cause diuresis.
  Other Names: Samsca
  Arms: Tolvaptan
Drug: Chlorothiazide — Chlorothiazide (Diuril) is an intravenous thiazide diuretic that works in the distal convoluted tubule of the nephron to cause diuresis.
  Other Names: Diuril
  Arms: Chlorothiazide
Drug: Metolazone — Metolazone (Zaroxolyn) is an oral thiazide diuretic that works in the distal convoluted tubule of the nephron to cause diuresis.
  Other Names: Zaroxolyn
  Arms: Metolazone

SUMMARY:
Broad Objectives: To determine the comparative efficacy of commonly employed strategies to overcome loop diuretic resistance when added to concomitant loop diuretics in hospitalized decompensated heart failure patients with hypervolemia

Specific Aims:

1. Compare the 48-hour weight change of either intravenous chlorothiazide or oral tolvaptan compared to standard-of-care oral metolazone when combined with standardized loop diuretic dosing for diuretic resistance in decompensated heart failure
2. Compare the adverse effects of electrolyte depletion and renal function changes between intravenous chlorothiazide or oral tolvaptan compared to standard-of-care oral metolazone when combined with standardized loop diuretic dosing for diuretic resistance in acute heart failure
3. Pharmacoeconomic analysis of the direct costs of intravenous chlorothiazide or oral tolvaptan compared to standard-of-care oral metolazone when combined with standardized loop diuretic dosing for diuretic resistance in acute heart failure

The investigators will conduct a dual center, randomized, double-blind, double-dummy, parallel design trial comparing: oral metolazone, intravenous chlorothiazide, or oral tolvaptan, in combination with loop diuretics in 60 patients hospitalized for hypervolemic decompensated heart failure and displaying loop diuretic resistance.

DETAILED DESCRIPTION:
Background:

The investigators aim to evaluate the optimal regimen for restoring diuretic efficacy in patients with decompensated heart failure demonstrating loop diuretic resistance, for which guideline-based recommendations are weak secondary to a lack of evidence. By comparing the efficacy, cost, and adverse effects of currently recommended therapies and testing a novel diuretic combination, the investigators will augment the dearth of data that exists regarding this clinical challenge.

Current heart failure guidelines recommend addition of a thiazide diuretic, listing either oral metolazone or intravenous chlorothiazide, to loop diuretic therapy as strategy to overcome loop diuretic resistance. At equipotent doses, these two therapies differ 250 fold in cost. To date, no prospective trial has compared the efficacy of these two commonly utilized therapies.

Tolvaptan, an oral vasopressin 2 receptor antagonist, could restore diuretic efficacy when used in combination with loop diuretics. While the safety of this combination has been established in the EVEREST trials, tolvaptan has been formally studied in a limited capacity as combination therapy to restore loop diuretic resistance. Hypokalemia is a common adverse effect of combining a thiazide and loop diuretic, increasing the risk of atrial and ventricular arrhythmias in a population who is already at high risk. Hypokalemia as not been reported with the combination of tolvaptan and loop diuretics, likely due to tolvaptan's distinctive mechanism of action. This potential benefit could provide tolvaptan a unique advantage for combination diuretic therapy in environments when electrolyte monitoring cannot be routinely performed or in patients with frequent arrhythmic events.

Methods:

All patients will provide informed consent prior to enrollment. All patients will be randomized in a 1:1:1 fashion using an electronic randomization tool embedded in REDCAP. All patients will be started on a 2L/day fluid restriction and a 2g/day sodium restriction. Decisions regarding the initiation, titration, or discontinuation of standard heart failure medications (Angiotensin Converting Enzyme Inhibitors, Angiotensin Receptor Blockers, Aldosterone Antagonists, Beta Blockers, digoxin, hydralazine, nitrates) are left to the discretion of the treating physicians. Patients will be randomized to either intravenous chlorothiazide 500mg IV Q12H + an oral placebo capsule Q12H or intravenous placebo infusion Q12H + a capsule containing either oral metolazone 5mg PO Q12H or oral tolvaptan 30mg once daily and placebo capsule in the evening dose. (Relative potency: Metolazone 100 fold more potent than chlorothiazide) All electrolyte repletion, loop diuretic dose titration, and concomitant therapies to enhance diuresis if needed will be utilized at the provider's discretion.

To prevent confounding heterogeneity in the diuretic treatment approach, a stepped care algorithm similar to the CARRESS-HF trial will be utilized for loop diuretics, both initial doses and subsequent dose changes, and for concomitant inotropes and vasodilators. A minimum furosemide equivalent dose of 580mg/24hrs (100mg IV bolus + 20mg/hr infusion rate) must be ordered at enrollment.

Outcomes The primary outcome will be 48-hour standing scale weight change (kg) from enrollment among the metolazone, intravenous chlorothiazide, and tolvaptan arms, using metolazone group as the comparator group for all other groups.

Secondary outcomes, using metolazone as the comparator group for each, will be:

* 48 hour net urine output (mls)
* mean change in serum creatinine,, blood urea nitrogen, and eGFR at 24 hours, 48hours, and at hospital discharge
* mean change in diuretic efficiency at 24 and 48 hours from baseline value at enrollment
* mean change in serum potassium at 24 and 48 hours from baseline value at enrollment
* mean change in serum sodium at 24 hours, 48hrs, and at discharge from baseline value at enrollment
* cumulative dose of potassium (mEq) and magnesium (g) supplementation administered at 24 and 48 hours
* incidence of severe hypokalemia
* need for escalation in study-directed loop diuretic therapy at 24 and 48 hours
* addition of vasoactive or inotropic medication at 24 and 48 hours
* Treatment failure (definition below)
* Patient-scored congestion visual analog scale score at baseline, 24 and 48 hours
* new cardiac arrhythmias (atrial and ventricular) during the study period
* receipt of inotropic therapy, dopamine, or nitroglycerin; requirement of ultrafiltration or hemodialysis during index hospitalization
* in-hospital mortality
* pharmacoeconomic analysis of the direct costs in each arm including the cost of: study medication, additional non-trial protocol laboratory analysis cost related to monitoring of electrolytes, treatment of study medication related adverse effects (arrhythmias, hypotension, electrolyte repletion), escalation of loop diuretic therapy doses, addition of additional therapies for suboptimal diuresis (inotropic therapy, vasodilators), and new initiation of renal replacement therapies (hemodialysis or ultrafiltration).

Study Definitions

* Urine output: Total urine volume (ml) from time of study enrollment to 48 hours
* Hypokalemia: Serum potassium value < 3.5mEq/L
* Severe Hypokalemia: Serum potassium value < 3.0mEq/L
* Hyponatremia: Serum sodium value < 135mEq/L
* Severe Hyponatremia: Serum sodium value < 130mEq/L and a decrease of 5mEq/L or more from enrollment serum sodium
* Overcorrection of serum sodium: increase in serum sodium from baseline by >12mEq/L in 24 hours, increase in >8mEq/L in 12 hours, or receipt of intravenous fluids because of symptoms of overcorrection of serum sodium regardless of the numerical rise
* Hypomagnesaemia : Serum magnesium value < 2mEq/L
* Diuretic efficiency = 24hr urine output/ 24hr Lasix equivalents in milligrams
* Weight: Standing weight on the same scale as used for baseline weight measurement
* New Atrial Arrhythmia: A "new" diagnosis of atrial arrhythmia (includes atrial fibrillation, atrial flutter, ectopic atrial tachycardia) lasting > 30 seconds OR any atrial arrhythmia which causes hemodynamic instability (MAP < 60 and requiring intervention)
* New Ventricular Arrhythmia: Ventricular tachycardia lasting longer than 30 seconds, or frequent non-sustained VT causing hemodynamic instability with MAP < 60 mmHg requiring intervention or > 1 intra-cardiac defibrillation or external cardiac defibrillation shock or ventricular fibrillation requiring defibrillation
* Hypotension: SBP < 85 for 2 repeated measurements within 30 minutes or lasting at least 30 minutes or symptomatic hypotension necessitating clinical intervention (defined as vasopressor support, intravenous fluid boluses, or initiation of inotropes)
* Treatment failure: Patients requiring additional non-study diuretic (spironolactone doses >75mg/day, eplerenone > 75mg/day, non-study thiazides (at a dose of metolazone 2.5mg or greater equivalence) or loop diuretics, or systemic acetazolamide (for diuretic indication), triamterene, or amiloride therapy) at any time during the 48-hour randomization period. These patients will be considered treatment failures for the purpose of analysis of the primary endpoint and all secondary endpoints.
* Patients whose cardiologist adds inotropic or vasodilator medications will not be considered treatment failures. Patients who require an increase in the loop diuretic regimen will also not be considered treatment failures.
* Medication costs will be defined as the Redbook average wholesale price at the time of the trial to reduce inter-institutional price differences and improve external validity of the analysis.

Statistical Analysis The investigators have collaborated with Department of Biostatistics at Vanderbilt University Medical Center to employ the best statistical methods that allow ther study to be realistic and achievable. Power calculations are difficult because of the lack of prospective trials comparing combination diuretic therapy and the numerous flaws in the methods of these previous studies. The investigators will utilize change in weight as the primary outcome because weight change has been utilized as a primary efficacy outcome in landmark heart failure diuretic trials (CARRESS-HF) and has less standard deviation than net urine output. In previous studies standard deviation of weight loss changes between groups varied with an approximate value of 1.6kg. If the minimum clinically meaningful difference in the experimental and control means is 1.5kg, the investigators will be able to reject the null hypothesis that the population means of the experimental and control groups are equal with 82.3% power. The Type I error probability associated with this test of this null hypothesis is 0.05. The investigators will utilize an intention-to-treat univariate Wilcoxon rank sum analysis for the independent continuous primary outcome variable using metolazone as the comparison group for both intravenous chlorothiazide and oral tolvaptan. The investigators will also perform a multivariate linear model adjusted analysis of the primary outcome to correct for baseline weight and loop diuretic regimen.

ELIGIBILITY:
Inclusion Criteria:

* age of 18 years or older
* hospital admission for hypervolemic decompensated heart failure complicated by loop diuretic resistance
* 24 hour telemetry monitoring on an inpatient ward
* basic metabolic panel laboratory assessment twice daily during the study period

Hypervolemia will be diagnosed by the admitting provider as either (i) pulmonary artery catheterization with a pulmonary capillary wedge pressure greater than 19mmHg plus a systemic physical exam finding of hypervolemia (peripheral edema, ascites, or pulmonary edema on auscultation) or (ii) in the absence of pulmonary artery catheterization data 2 of the following signs or symptoms: peripheral edema ascites, jugular venous pressure > 10mmHg, or pulmonary edema on chest x-ray.

Loop diuretic resistance is defined as a provider decision to pursue combination diuretic therapy because of failure to reach provider defined adequate diuresis (can not exceed urine output of 2 L in past 12 hours) despite receipt of an intravenous loop diuretic dose of a furosemide equivalent of at least 240mg/day over at least the past 12 hours (40mg furosemide = 20mg torsemide = 1mg bumetanide).

Exclusion Criteria:

* decision to pursue hemodialysis by a nephrologist
* estimated glomerular filtration rate by the MDRD equation < 15ml/min/m2
* systolic blood pressure < 85mmHg
* pregnancy
* serum potassium < 3.0mEq/L
* serum sodium > 145mEq/L or < 130mEq/L
* severe malnutrition
* advanced liver disease
* inability to perform standing weights
* inability to collect and measure urine with either a foley catheter or urine collection containers
* concomitant therapy with strong CYP3A4 inhibitors/inducers (systemic ketoconazole, clarithromycin, itraconazole, telithromycin, saquinavir, nelfinavir, ritonavir, nefazodone, rifampin, rifabutin, rifapentine, phenytoin, phenobarbital, carbamazepine, St. John's Wort)
* concomitant therapy with p-glycoprotein inhibitors (cyclosporine, erythromycin, tacrolimus, dronedarone, quinidine, or verapamil)
* non-study diuretics (spironolactone doses >75mg/day, eplerenone > 75mg/day, non-study thiazides or loop diuretics, or systemic acetazolamide, triamterene, or amiloride therapy)
* thiazides administration in the previous 24 hours prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02; Primary Completion 2018-09-27 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zachary L Cox, PharmD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Cox ZL, Hung R, Lenihan DJ, Testani JM. Diuretic Strategies for Loop Diuretic Resistance in Acute Heart Failure: The 3T Trial. JACC Heart Fail. 2020 Mar;8(3):157-168. doi: 10.1016/j.jchf.2019.09.012. Epub 2019 Dec 11. PMID 31838029

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metolazone | Chlorothiazide | Tolvaptan
Started | 20 | 20 | 20
Completed | 15 | 18 | 20
Not Completed | 5 | 2 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Protocol Violation | 2 | 1 | 0
Not completed — Physician Decision | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metolazone | Chlorothiazide | Tolvaptan | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (15) | 67 (11) | 58 (14) | 62 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 8 | 17
  Male | 15 | 16 | 12 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 13 | 12 | 15 | 40
  Black | 6 | 8 | 5 | 19
  Other | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 60
Number of Patients with HF reduced Ejection fraction [Count of Participants; unit: Participants] | 12 | 16 | 18 | 46
Number of Patients with HF preserved Ejection fraction [Count of Participants; unit: Participants] | 8 | 4 | 2 | 14
Ischemic cardiomyopathy [Count of Participants; unit: Participants] | 6 | 9 | 8 | 23
Mean Left ventricular ejection fraction (%) [Mean (Standard Deviation); unit: %] | 35 (19) | 29 (17) | 27 (13) | 30 (16)
Number of patients with coronary artery disease [Count of Participants; unit: Participants] | 10 | 12 | 13 | 35
Number of patients with hypertension [Count of Participants; unit: Participants] | 18 | 18 | 13 | 49
Number of patients with diabetes mellitus [Count of Participants; unit: Participants] | 12 | 19 | 11 | 42
Number of patients with chronic kidney disease [Count of Participants; unit: Participants] | 16 | 16 | 12 | 44
Number of patients with atrial fibrillation [Count of Participants; unit: Participants] | 13 | 10 | 9 | 32
Cumulative IV Loop diuretic dose in Furosemide Equivalents for previous 24 hours (mg/24 hrs) [Mean (Standard Deviation); unit: mg/24 hours] | 680 (517) | 611 (464) | 546 (324) | 612 (429)
Total urine output in past 12 hours (mls) [Mean (Standard Deviation); unit: ml] | 1170 (412) | 1372 (500) | 1022 (465) | 1118 (476)
Diuretic Efficiency [Mean (Standard Deviation); unit: ml urine output/ 40mg IV furosemide] | 199 (129) | 254 (161) | 174 (96) | 209 (134)
Serum sodium (mEq/L) [Mean (Standard Deviation); unit: mEq/L] | 139 (2) | 138 (4) | 137 (3) | 138 (3)
Serum potassium (mEq/L) [Mean (Standard Deviation); unit: mEq/L] | 3.9 (0.5) | 4.0 (0.4) | 4.0 (0.5) | 3.9 (0.5)
Serum chloride (mEq/L) [Mean (Standard Deviation); unit: mEq/L] | 100 (6) | 100 (4) | 100 (5) | 100 (5)
BUN (mg/dl) [Mean (Standard Deviation); unit: mg/dl] | 46 (19) | 48 (31) | 41 (23) | 45 (25)
Serum Creatinine (mg/dl) [Mean (Standard Deviation); unit: mg/dl] | 2.0 (0.9) | 2.1 (0.7) | 1.8 (0.7) | 1.9 (0.7)
Glomerular filtration rate (ml/min/m2) [Mean (Standard Deviation); unit: ml/min/m2] | 41 (19) | 36 (15) | 46 (24) | 41 (20)
Systolic blood pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] | 114 (13) | 119 (20) | 114 (12) | 115 (15)
Patient-Reported Visual Analog Congestion Score from 0 cm (worst symptoms) to 10cm (best) [Mean (Standard Deviation); unit: cm on dyspnea analog scale] | 2.5 (2.2) | 4.1 (2.2) | 3.8 (2.3) | 3.4 (2.3)
Number of patients on Beta blocker therapy [Count of Participants; unit: Participants] | 16 | 13 | 17 | 46
Number of patients on ACEI/ARB/ARNI therapy [Count of Participants; unit: Participants] — ACEI= angiotensin converting enzyme inhibitor; ARB = angiotensin receptor blocker; ARNI = angiotensin receptor-neprilysin inhibitor
  Participants | 6 | 6 | 9 | 21
Number of patients on Aldosterone antagonist therapy [Count of Participants; unit: Participants] | 10 | 6 | 11 | 27
Number of patients on Intravenous Inotrope therapy [Count of Participants; unit: Participants] | 2 | 2 | 2 | 6
Number of patients on Loop diuretic infusion 100mg bolus & 20mg/h [Count of Participants; unit: Participants] | 10 | 10 | 9 | 29
Number of patients on Loop diuretic infusion 100mg bolus & 30mg/h [Count of Participants; unit: Participants] | 10 | 10 | 11 | 31

OUTCOME MEASURES:

1. Primary Outcome: Weight Change Over 48 Hours
Description: The primary outcome will be 48-hour standing scale weight change (kg) from enrollment among the metolazone, intravenous chlorothiazide, and tolvaptan arms, using metolazone group as the comparator group for all other groups.
Time Frame: 48 hours
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Metolazone | Chlorothiazide | Tolvaptan
Number analyzed (Participants) | 20 | 20 | 20
kg | -4.6 (2.7) | -5.8 (2.7) | -4.1 (3.3)

2. Secondary Outcome: Net Urine Output
Description: Net urine output from enrollment to the end of study at 48 hours measured in liters
Time Frame: 48 hours
Population: Intention to treat
Measure: Median (Inter-Quartile Range); unit: liters
Arm/Group | Metolazone | Chlorothiazide | Tolvaptan
Number analyzed (Participants) | 20 | 20 | 20
liters | -7.8 [-10.1 to -6.6] | -8.8 [-10.9 to -7.4] | -9.8 [-13.8 to -6.4]

3. Secondary Outcome: Mean Change in Serum Creatinine
Description: Mean change in serum creatinine (mg/dl) from enrollment to end of study at 48 hours
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Metolazone | Chlorothiazide | Tolvaptan
Number analyzed (Participants) | 20 | 20 | 20
mg/dl | 0.3 (0.3) | 0.5 (0.5) | 0.03 (0.3)

4. Secondary Outcome: Mean Change in Glomerular Filtration Rate at Discharge
Description: Mean change in glomerular filtration rate from enrollment to end of study at hospital discharge, an average of 5 days
Time Frame: hospital discharge an average of 5 days
Measure: Mean (Standard Deviation); unit: ml/min/m2
Arm/Group | Metolazone | Chlorothiazide | Tolvaptan
Number analyzed (Participants) | 20 | 20 | 20
ml/min/m2 | -2 (19) | -2 (13) | -6 (10)

5. Secondary Outcome: Mean Change in Serum Potassium
Description: Mean change in serum potassium (mEq/L) from enrollment to end of study at 48 hours
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Metolazone | Chlorothiazide | Tolvaptan
Number analyzed (Participants) | 20 | 20 | 20
mEq/L | -0.1 (0.7) | -0.2 (0.5) | 0.1 (0.5)

6. Secondary Outcome: Potassium Supplementation
Description: Cumulative dose of potassium supplementation (mEq) administered from enrollment to end of study at 48 hours
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: mEq
Arm/Group | Metolazone | Chlorothiazide | Tolvaptan
Number analyzed (Participants) | 20 | 20 | 20
mEq | 103 (131) | 63 (60) | 58 (56)

7. Secondary Outcome: Number of Patients With Hypokalemia
Description: Incidence of hypokalemia (serum potassium less than 3.5mEq/L ) from enrollment to end of study
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Metolazone | Chlorothiazide | Tolvaptan
Number analyzed (Participants) | 20 | 20 | 20
Participants | 3 | 2 | 2

8. Secondary Outcome: Number of Patients With Escalation of Loop Diuretic Therapy
Description: Provider escalation of loop diuretic dosage at 24 hours for urine output less than 3 L at 24 hours
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Metolazone | Chlorothiazide | Tolvaptan
Number analyzed (Participants) | 20 | 20 | 20
Participants | 4 | 4 | 2

9. Secondary Outcome: Number of Patients With Cardiac Arrhythmias
Description: Incidence of new atrial or ventricular arrhythmias from enrollment to end of study at 48 hours
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Metolazone | Chlorothiazide | Tolvaptan
Number analyzed (Participants) | 20 | 20 | 20
Participants | 0 | 0 | 0

10. Secondary Outcome: Number of Patients With Symptomatic Hypotension
Description: SBP < 85 mmHg plus medical intervention for symptomatic hypotension
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Metolazone | Chlorothiazide | Tolvaptan
Number analyzed (Participants) | 20 | 20 | 20
Participants | 2 | 0 | 2

11. Secondary Outcome: Change in eGFR From Baseline to 48 Hours
Description: Change in estimated glomerular filtration rate (ml/min/m2) from baseline to 48 hours
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: ml/min/m2
Arm/Group | Metolazone | Chlorothiazide | Tolvaptan
Number analyzed (Participants) | 20 | 20 | 20
ml/min/m2 | -6 (7) | -9 (9) | 2 (11)

12. Secondary Outcome: Mean Change in Serum Sodium
Description: Mean change in serum sodium (mEq/L) from enrollment to end of study at 48 hours
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Metolazone | Chlorothiazide | Tolvaptan
Number analyzed (Participants) | 20 | 20 | 20
mEq/L | -1 (3) | -1 (3) | 4 (5)

13. Other Pre Specified Outcome: Number of Patients With In-hospital Mortality
Description: Incidence of death from study enrollment to hospital discharge, an average of 5 days
Time Frame: Enrollment to hospital discharge an average of 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Metolazone | Chlorothiazide | Tolvaptan
Number analyzed (Participants) | 20 | 20 | 20
Participants | 0 | 0 | 0

14. Other Pre Specified Outcome: Number of Patients With New Inotrope Utilization
Description: Incidence of new initiation of dopamine, dobutamine, or milrinone from enrollment to end of study at 48 hours
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Metolazone | Chlorothiazide | Tolvaptan
Number analyzed (Participants) | 20 | 20 | 20
Participants | 1 | 0 | 2

15. Other Pre Specified Outcome: Number of Patients With Renal Replacement Therapy Utilization
Description: Incidence of Renal replacement therapy utilization (hemodialysis, ultrafiltration) from enrollment to hospital discharge, an average of 5 days
Time Frame: enrollment to hospital discharge an average of 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Metolazone | Chlorothiazide | Tolvaptan
Number analyzed (Participants) | 20 | 20 | 20
Participants | 0 | 0 | 0

16. Other Pre Specified Outcome: Diuretic Efficiency
Description: Diuretic Efficiency is calculated as 48hr urine output/ 48hr Furosemide equivalents in milligrams
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: UOP / 40mg IV furosemide
Arm/Group | Metolazone | Chlorothiazide | Tolvaptan
Number analyzed (Participants) | 20 | 20 | 20
UOP / 40mg IV furosemide | 217 (107) | 294 (123) | 326 (213)

17. Other Pre Specified Outcome: Change in Serum Chloride From Baseline
Description: Change in serum chloride (mEq/L) from baseline to 48 hrs
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Metolazone | Chlorothiazide | Tolvaptan
Number analyzed (Participants) | 20 | 20 | 20
mEq/L | -7 (4) | -7 (2) | 2 (3)

18. Other Pre Specified Outcome: Change in Patient Congestion Score
Description: Participants will score their congestion on a 10cm scale ranging from "Best" (10cm) to "Worst" (0cm). Change in score (units in centimeters) from baseline to 48 hours.
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: cm of dyspena analog scale
Arm/Group | Metolazone | Chlorothiazide | Tolvaptan
Number analyzed (Participants) | 20 | 20 | 20
cm of dyspena analog scale | 4.0 [2.5 to 7.0] | 3.0 [2.0 to 4.6] | 3.0 [2.0 to 5.0]

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 48 hour study and over a subsequent 30 day follow up period. Events detailed below are through the 30 day follow up period.
Arm/Group | Metolazone | Chlorothiazide | Tolvaptan
All-Cause Mortality (participants affected / at risk) | 0/20 | 1/20 | 1/20
Serious Adverse Events (participants affected / at risk) | 2/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 5/20 | 6/20 | 10/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metolazone (N=20) | Chlorothiazide (N=20) | Tolvaptan (N=20)
Hypotension (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) — Severe, symptomatic hypotension (SBP < 85 mmHg) requiring study drug discontinuation and medical intervention.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metolazone (N=20) | Chlorothiazide (N=20) | Tolvaptan (N=20)
Increase in serum sodium (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) — Rapid increases in serum sodium
Non-severe hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) — transient symptomatic hypotension not requiring study drug discontinuation
Gout flare (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) — symptomatic gout attack
muscle cramping (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1)
Serum creatinine increase > 1mg /dl (Renal and urinary disorders) | 1 (1) | 3 (3) | 0 (0)
Severe Hypokalemia < 3.0 mEq/L (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea/vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Delirium (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
cardioembolic stroke (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
We conducted a single-center trial. We were not powered for non-inferiority. The observed weight loss standard deviation exceeded the expected standard deviation, reducing power. Outcomes at discharge were influenced by open-label diuretic therapy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-08-31): https://cdn.clinicaltrials.gov/large-docs/53/NCT02606253/Prot_SAP_ICF_000.pdf